CLINICAL TRIAL: NCT00340730
Title: Community Based Youth Injury Prevention Program
Status: Completed | Type: Observational
Sponsor: Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999902070; 02-CH-N070
Record Dates: First submitted 2006-06-19; First posted 2006-06-21 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2006-11-02

CONDITIONS: Violence; Intervention
Keywords: Health Education; Mentoring; Parenting; Social Skills Training; Violence; Intervention; Youth Injury
MeSH Terms: conditions — Health Education

SUMMARY:
America's greatest resource is its youth, but that resource is increasingly threatened by violence. Recommendations for violence prevention have highlighted the need to focus on youth and to explore targeted interventions Nowhere is the need greater than in our nation's capital where the intentional injury fatality rate for youth age 14-19 is higher than any of the 50 states. This study builds on the CDC-supported project Adolescent Violence: A Community-Based Strategy which instituted citywide surveillance on injuries, conducted by researchers at the Children's National Medical Center. In this study, the same researchers will extend that work by testing an individualized intervention to reduce violent behavior among a sample of assault-injured youth, age 9-15, who present at the Emergency department (ED). 196 youths and their families will be included in this randomized trial, with 98 families assigned to the individualized intervention condition and 98 families assigned to the control condition. Families will be followed for 18 months. To address issues of attrition over the 18 months that the study follows, approximately twice as many families, or 400 families, will be recruited to participate in the study.

DETAILED DESCRIPTION:
America's greatest resource is its youth, but that resource is increasingly threatened by violence. Recommendations for violence prevention have highlighted the need to focus on youth and to explore targeted interventions. Nowhere is the need greater than in our nation's capital where the intentional injury fatality rate for youth age 14-19 is higher than any of the 50 states. This study builds on the CDC-supported project Adolescent Violence: A Community-Based Strategy which instituted citywide surveillance on injuries, conducted by researchers at the Children's National Medical Center. In this study, the same researchers will extend that work by testing an individualized intervention to reduce violent behavior among a sample of assault-injured youth, age 9-15, who present at the Emergency Department (ED). 196 youths and their families will be included in this randomized trial, with 98 families assigned to the individualized intervention condition and 98 families assigned to the control condition. Families will be followed for 18 months. To address issues of attrition over the 18 months that the study follows, approximately twice as many families, or 400 families, will be recruited to participate in the study.

ELIGIBILITY:
* INCLUSION CRITERIA:

A consecutive sample of youth presenting to the ED or hospitalized for interpersonal assault injuries meeting the following criteria will be recruited: Interpersonal injuries; Youth age 9-15 and their parents or guardians.

Youth and their families will be excluded from participation for the following reasons: Injuries due to child abuse and sexual abuse; those with severe psychopathology (i.e., severe depression or psychosis s measured by extreme responses on selected CBCL questions); Youth or their parents with an inability to comprehend questions for reasons of cognitive ability or language will be excluded.

Min Age: 7 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 392
Dates: Start 2001-12-04; Study Completion 2006-11-02

CONTACTS AND LOCATIONS:
Locations (1):
- National Institute of Child Health and Human Development (NICHD), Bethesda, Maryland, United States

REFERENCES:
- [Background] Fingerhut LA, Ingram DD, Feldman JJ. Firearm homicide among black teenage males in metropolitan counties. Comparison of death rates in two periods, 1983 through 1985 and 1987 through 1989. JAMA. 1992 Jun 10;267(22):3054-8. PMID 1514955